CLINICAL TRIAL: NCT04916080
Title: N-acetyl Cysteine: the Effectiveness and Safety in a Cohort of Pediatric Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Mostafa Ahmed, Assistant professor, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMBSUREC. FWA00015574
Record Dates: First submitted 2021-04-30; First posted 2021-06-07 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: 50 children with chronic kidney disease will be assessed for iron profile, oxidative stress status and left ventricular functions before and after treatment with N-acetyl cysteine for 3 months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- after treatment (Experimental): chronic kidney disease patients after receiving NAC for 3 months
  Interventions: Drug: N-acetyl cysteine

INTERVENTIONS:
Drug: N-acetyl cysteine — mucolytic and anti-oxidant. Dose 10mg/Kg/ 12 hours orally
  Other Names: NAC

SUMMARY:
Anemia is a common comorbidity of CKD and is associated with a decreased quality of life and increased healthcare resource utilization. Anemia increases the risk of CKD progression, cardiovascular complications, and overall mortality. The current standard of care includes oral or intravenous iron supplementation, erythropoiesis-stimulating agents, and red blood cell transfusion. Treatment with high doses of erythropoiesis-stimulating agents increases rates of hospitalization, cardiovascular events, and mortality. Resistance to erythropoiesis-stimulating agents is a therapeutic challenge in many patients .

NAC reduces the risk of progression of CKD of any etiology to end stage renal disease (ESRD) but the mechanism by which it reduces the progression of CKD to ESRD is unclear. It may be because of its antioxidant and vasodilatory nature. Prolonged duration of administration and higher dosage of NAC can protect kidneys.

DETAILED DESCRIPTION:
All patients with chronic kidney disease on regular hemodialysis will be enrolled.

- Study location: The patients will be recruited from pediatric nephrology department, Cairo University Children's Hospital and Beni Suef University.

History taking including the age, sex, primary cause of CKD, onset of hemodialysis, medications including erythropoietin dose, frequency, and duration, oral or intravenous iron therapy, and frequency of blood transfusion.

Clinical examination focusing on pallor, blood pressure, and anthropometric measurements and their percentile.

Investigations including hemoglobin level at the start of the study and every month during the study period, serum ferritin, alanine aminotransferase, total oxidative stress (TOS), total antioxidant capacity (TAC), and oxidative stress index (OSI) at the start and after 3 months of the onset of the study.

Patients will receive N-acetyl cysteine (10 mg/kg/day, orally). The duration of the study will 3 months.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients with chronic kidney diseases stage 3, 4 or 5

Exclusion Criteria:

* Unwilling to participate in the study.
* non-compliant patients on the standard care of CKD.

  * Patients with cardiac, endocrinal, and hepatic complications.
  * Asthma or known allergy to NAC.
  * Any chronic infections prior to or during the study period.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
hemoglobin (gm%) | 3 months
  the change in levels of hemoglobin after treatment
oxidative status | 3 months
  rate of change of total oxidative status after treatment using ELISA kits
left ventricular function | 3 months
  rate of change of left ventricular functions before and after treatment by electrocardiography
serum Ferritin level (mg/dl) | 3 months
  the change in levels of d ferritin after treatment using specific kits
Anti-oxidative status | 3 months
  rate of change of anti oxidant capacity after treatment

SECONDARY OUTCOMES:
serious side effects | 3 months
  elevation of ALT levels

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Beni-Suef university hospital, Banī Suwayf
  - Pediatric nephrology and transplantation unite.Aboelrish children hospital, Cairo